CLINICAL TRIAL: NCT05896839
Title: A Phase 2 Study of Nivolumab and Ipilimumab in Combination With Sirolimus and Prednisone in Kidney Transplant Recipients With Selected Unresectable or Metastatic Cutaneous Cancers
Brief Title: Immunotherapy in Combination With Prednisone and Sirolimus for Kidney Transplant Recipients With Unresectable or Metastatic Skin Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-04306; NCI-2023-04306 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ETCTN10614; 10614 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10614 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2023-06-08; First posted 2023-06-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8; Metastatic Basal Cell Carcinoma; Metastatic Carcinoma in the Skin; Metastatic Melanoma; Metastatic Merkel Cell Carcinoma; Metastatic Skin Squamous Cell Carcinoma; Unresectable Basal Cell Carcinoma; Unresectable Melanoma; Unresectable Merkel Cell Carcinoma; Unresectable Skin Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Melanoma; Carcinoma, Merkel Cell | interventions — Biopsy; Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab; Prednisone; deltacortene; prednylidene; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nivolumab and ipilimumab) (Experimental): See detailed description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Kidney Biopsy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Prednisone; Drug: Sirolimus

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Kidney Biopsy — Undergo kidney biopsy
  Other Names: Biopsy of Kidney; Renal Biopsy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Sirolimus — Given PO
  Other Names: AY 22989; AY-22989; AY22989; RAPA; Rapamune; Rapamycin; SILA 9268A; SILA-9268A; SILA9268A; WY 090217; WY-090217; WY090217

SUMMARY:
This phase II trial tests the combination of nivolumab and ipilimumab with sirolimus and prednisone for the treatment of skin (cutaneous) cancer that cannot be removed by surgery (unresectable) or that has spread from where it first started to other places in the body (metastatic) in kidney transplant recipients. Immunotherapy with nivolumab and ipilimumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Sirolimus and prednisone are immunosuppressants that are given to keep the body from rejecting the transplanted kidney. Giving nivolumab and ipilimumab in combination with sirolimus and prednisone may kill more cancer cells, while also keeping the transplanted kidney healthy, in patients with unresectable or metastatic cutaneous cancer who have received a kidney transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of kidney transplant recipients with selected advanced cutaneous cancers who at 14 weeks after administration of prednisone, sirolimus, nivolumab, and ipilimumab experience complete response (CR), partial response (PR), or stable disease (SD) without allograft loss.

SECONDARY OBJECTIVE:

I. To estimate the objective response rate (ORR), rate of allograft loss, and durations of progression-free survival (PFS) and overall survival (OS) in the study population.

EXPLORATORY OBJECTIVES:

I. To characterize correlates of the host immune response including, but not limited to:

Ia. Histopathological characteristics of allograft rejection/loss; Ib. Immunological changes in the tumor microenvironment (e.g., changes in T-cell subset populations or expression of immune checkpoint molecules) in paired biopsies obtained pre-treatment and on-treatment; Ic. Characteristics of anti-programmed death-1 (PD-1)-associated immune-mediated adverse reactions (IMARs) in this patient population treated with immunosuppression; Id. To identify upregulated immune-related genes using multiplex quantitative reverse transcription polymerase chain reaction (qRT-PCR).

II. To observe whether changes in donor-derived cell-free deoxyribonucleic acid (DNA) (dd-cfDNA) as a marker for allograft rejection.

III. To compare baseline patient allograft/donor characteristics, to include human leukocyte antigen (HLA) status, date of transplant, presence of donor specific antibodies, history of prior rejection, and Calculated Panel Reactive Antibodies score, in patients who experience and do not experience rejection while on this study.

IV. To observe the objective response rate (ORR) of patients who achieve PR/CR or stable disease for >= 6 months with eventual progressive disease requiring re-induction with nivolumab + ipilimumab (receive > 4 doses of nivolumab + ipilimumab).

OUTLINE:

Patients receive sirolimus orally (PO) and prednisone PO daily, starting 7 days prior to cycle 1 day 1 of immunotherapy. Patients also receive nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 8 of cycle 1 and day 1 of cycle 2. Six weeks after the first dose of nivolumab and ipilimumab, patients undergo tumor response assessment. Patients who achieve stable disease (SD), partial response (PR), or complete response (CR) receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for a total of 24 cycles in the absence of disease progression or unacceptable toxicity. Patients who had disease progression at this time or any time on trial may receive nivolumab IV and ipilimumab IV on day 1 of each cycle. Cycles repeat every 3 weeks for 2 cycles, in the absence of unacceptable toxicity. Patients are then assessed for tumor response again after 6 weeks and receive nivolumab monotherapy if they achieve SD, PR, or CR. If patients have progressive disease, they may receive nivolumab monotherapy or discontinue study treatment.

Patients may undergo magnetic resonance imaging (MRI) during screening, undergo tumor biopsy on study and undergo computed tomography (CT) scan and blood sample collection throughout the study. Patients may undergo kidney biopsy if rejection is suspected.

Patients follow up every 12 weeks for 1 year after stopping therapy, then every 16 weeks for the second year after stopping and then every 20 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be kidney transplant recipients with a functioning allograft who do not currently require dialysis
* Patient's age must be >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of nivolumab and ipilimumab in kidney transplant recipients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials
* Patients must have histologically or cytologically confirmed non-uveal melanoma, basal cell carcinoma, Merkel cell carcinoma, or cutaneous squamous cell carcinoma for which standard non-immunological medical, surgical, or radiation therapy would be insufficient (i.e., patients who are not surgical candidates). Patients with cutaneous squamous cell carcinoma or Merkel cell carcinoma may enroll without prior medical therapy (e.g., cetuximab or chemotherapy respectively). Non-immunologic standard therapies that patients must have received, refused or for which patients were ineligible include:

  * For patients with BRAF-mutant melanoma, prior therapies include BRAF/MEK inhibitors
  * For patients with Basal cell carcinoma, prior therapies include hedgehog pathway inhibitors
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, i.e., at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm by chest x-ray or as >= 10 mm with CT scan, magnetic resonance imaging (MRI), or calipers by clinical exam is preferred, but not required
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%) performance status criteria
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 50,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine =< 3 x ULN
* dd-cfDNA =< 1.0% and =< 61% increase
* The effects of nivolumab and ipilimumab on the developing human fetus are unknown. For this reason, and because other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential (WOCBP) receiving nivolumab must continue contraception for a period of 5 months after the last dose of nivolumab. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [B-HCG]) during the screening period. Follow-up evaluations will include interval sexual/menstrual histories as needed.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately.

WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. Women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL to be considered postmenopausal.

* Human immunodeficiency virus (HIV)-infected patients will be eligible for this trial if they are on effective antiretroviral regimens utilizing non-CYP-interactive agents and have an undetectable viral load. If there is evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy, if indicated. If there is history of hepatitis C virus (HCV) infection, the patient must have been treated and have undetectable HCV viral load.
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have received a liver, lung, heart, or pancreas transplant; or allogeneic stem cell transplant; or any kind of bone marrow transplant
* Patients unwilling or unable to undergo dialysis in the event of allograft failure
* Patients with prior evidence of human leukocyte antigen (HLA) or non-HLA donor-specific antibodies (DSA)
* Patients with a history of antibody- or cell-mediated allograft rejection within 3 months of study entry
* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment
* Patients may have received prior anti-PD-(L)1 therapy; however, patients must not have any other checkpoint antibody targeting T-cell co-stimulation within 1 year of study enrollment. Prior history of adjuvant therapy is allowed if received over 1 year prior to enrollment. Prior receipt of oncolytic therapy (e.g., TVEC, RP1) is allowed
* Patients must not be receiving any other investigational agents
* Patients with leptomeningeal metastases, more than 3 untreated central nervous system (CNS) metastases, untreated brain metastases measuring >1cm, or requiring treatment-dose steroids (> 10 mg/day prednisone equivalents) for CNS-related symptoms. Exclusions are due to concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other AEs. Patients with brain metastases meeting the above requirements are permitted to enroll
* Patients must not have a history of severe hypersensitivity reaction to any monoclonal antibody
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in the study
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other significant condition(s) that would make this protocol unreasonably hazardous
* Pregnant women are excluded from this study because nivolumab and ipilimumab have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with nivolumab or ipilimumab. These potential risks may also apply to other agents used in this study
* Patients with autoimmune disease that is active or might recur and affect vital organ function will be eligible only after consultation with the study PI. Guillain-Barre (GB) syndrome, bullous skin disease, Stevens Johnson syndrome, or toxic epidermal necrolysis will be excluded
* Patients must not have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study. In addition, patients with a history of cardiac disease including coronary artery disease (CAD), myocardial infarction (MI), cardiomyopathy, arrhythmia, heart block, should have an evaluation by history pulmonary embolism (PE) and appropriate testing to allow evaluation of any events that may occur on study. These may include troponin, electrocardiogram (EKG), echocardiogram (ECHO) as clinically indicated and may include results already in the medical record if available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease control without allograft loss | At 14 weeks
  Defined as complete or partial response (CR; PR) or stable disease (SD), at 14 weeks per response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The percent of kidney transplant recipients who experience CR/PR/SD at 14 weeks and do not experience allograft loss after administration of nivolumab, ipilimumab, sirolimus, and prednisone will be calculated, along with the corresponding exact 95% confidence interval (CI).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  Defined as the proportion of subjects whose best overall response from baseline is either a CR or PR, based on RECIST 1.1 criteria. ORR will be estimated along with 95% exact CI.
Rate of allograft loss and rejection | Up to 5 years
  Renal allograft rejection rate will be estimated as the proportion of subjects who experience markers of allograft rejection. Allograft loss is defined as allograft rejection leading to complete, permanent, and irreversible loss-of-function of the renal allograft.
Duration of response (DOR) among patients who experience CR or PR | From the time criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent disease or PD is documented, up to 5 years
  DOR will be summarized using the Kaplan-Meier method.
Progression-free survival (PFS) | From the first dose of nivolumab + ipilimumab to the date of the first documented tumor progression or death due to any cause, whichever occurs first, up to 5 years
  Kaplan-Meier curves will be used to summarize PFS.
Overall survival | From the first dose of nivolumab + ipilimumab to the date of death from any cause, up to 5 years
  Kaplan-Meier curves will be used to summarize OS.

CONTACTS AND LOCATIONS:
Overall Officials: Evan J Lipson, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (26):
- United States (26):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm